CLINICAL TRIAL: NCT02437942
Title: An Examination of the Anatomical and Biomechanical Diagnoses That Exist in Athletic Groin Pain Patients and the Effects of a Biomechanics Led Rehabilitation Intervention in These Same Patients
Brief Title: Anatomical, Radiological and Biomechanical Examination of Athletic Groin Pain Patients and Physical Therapy Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sports Surgery Clinic, Santry, Dublin (Other)
Collaborators: Insight Centre for Data Analytics (Other); Science Foundation Ireland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSC-Groin-001
Record Dates: First submitted 2015-04-29; First posted 2015-05-08 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Groin Pain
Keywords: Athletic injuries; chronic; rehabilitation; diagnosis; biomechanics
MeSH Terms: conditions — Athletic Injuries; Bronchiolitis Obliterans Syndrome; Disease

ARMS (1):
- Biomechanics led physical therapy rehabilitation (Experimental): Physical therapy exercise rehabilitation
  Interventions: Other: Biomechanics led physical therapy rehabilitation

INTERVENTIONS:
Other: Biomechanics led physical therapy rehabilitation — Rehabilitation intervention will consist of movement control (3 days per week), whole body strength and power (2 days per week), linear running mechanics (3 days per week), multi-directional mechanics (3 days per week), conditioning sessions (2 days per week). Rehabilitation will continue until physical therapist deems the athlete ready to return to sport.

SUMMARY:
Athletic groin pain (AGP) is a chronic condition common in multi-directional sports (Walden et al. 2007, Robinson et al. 2004, Murphy et al. 2012). It is a complex injury with a challenging diagnosis. Dramatic differences in the anatomical diagnoses of AGP cohorts exist in the literature (Renstrom et al. 1980, Lovell et al. 1995, Holmich et al. 2007, Bradshaw et al. 2008). This may be due to the complexity of the anatomy in the region and the absence of magnetic resonance imaging (MAGNETIC RESONANCE IMAGE) to confirm clinical examination.

Dynamic actions undertaken in field sports (including change of direction cutting) are particularly associated with the development of athletic groin pain (Holmich et al. 2014). Dynamic multi-plane, multi-joint actions can overload musculoskeletal and fascial structures in the hip and groin. Despite this, traditional groin pain assessments do not involve an examination of sport specific actions. An examination of jumping, hopping and cutting mechanics, which is possible with the use of three dimensional motion capture techniques, will provide additional information with which to diagnosis and rehabilitate athletes.

While the majority of published studies on AGP have focused on surgical management (Serner et al. 2015), exercise therapy has been found to be an effective treatment (Holmich et al. 1995). In exercise therapy studies the best results were shown by Holmich et al (1995) where subjects suffered for an average of 9.9 months with symptoms and a strength and stability program focused on adductor strength returned them to sport in 18.5 weeks. The latest paper on rehabilitation by Jardi et al. demonstrates little improvement with a mean time to return to training of 86 days +/-15. The focus remains on improving strength of isolated muscle groups and not attempting to address underlying biomechanical abnormalities that may be leading to overload. Accurate biomechanical assessment and individualized rehabilitation based on the high speed multiplanar movements that drive the athlete's symptoms may enhance the efficiency of rehabilitation. Moreover post-rehabilitation changes in biomechanical factors may provide a further insight into the biomechanical factors associated with AGP.

The purpose of this study was to:

1. Describe clinical presentation (physical examination and magnetic resonance imaging findings) for a group of athletes presenting with AGP
2. To describe the different biomechanical diagnoses that exist in AGP patients
3. To examine the effects of a biomechanics led exercise intervention to rehabilitate chronic groin pain

It is hypothesised that standardised magnetic resonance imaging will aid in the anatomical diagnosis of athletic groin pain patients. From a biomechanics perspective, distinct subgroups/clusters will exist that differ from each other in how they undertake dynamic sport specific actions. These distinct clusters will describe potential biomechanical diagnoses that exist in groin pain patients. A biomechanics led rehabilitation program will return groin pain patients back to sport more quickly than previous rehabilitation programs without biomechanical diagnostic information.

Brief protocol Participants will be recruited from patients with chronic athletic groin pain who present for investigation and rehabilitation at Sports Surgery Clinic, Ireland. A standardised clinical examination will be undertaken including range of motion assessment, pain provocation and load tolerance tests, and palpation.

A Magnetic Resonance Image of the hip and groin region will then be undertaken and read by a consultant sports physician.

Biomechanical assessment will include capturing of jumping, hopping and cutting mechanics through the use of three dimensional motion capture technology and force plates. Here reflective markers are placed on the skin at anatomical landmarks. These markers are picked up by the cameras and tracked at 200 frames per second. Participants will contact the force plate with their foot on undertaking the movements. Force and marker data will be combined to calculate joint angles and moments.

Physical therapy assessment will include an assessment of functional movement, range of motion testing, adductor squeeze tests, strength assessment of hip and trunk. Physiotherapists will utilise three dimensional biomechanical data during cutting and landing to inform individualised rehabilitation. Rehabilitation will consist of movement control, whole body strength and power, linear running mechanics, multi-directional mechanics and conditioning sessions. Participants will have follow up physical therapy appointments approximately every two weeks. A hip and groin outcome score (HAGOS) will be used to monitor the morbidity and severity of the injury throughout the rehabilitation process.

Once the physiotherapist determines that the patient is ready to return to play a biomechanical re-test will be undertaken.

DETAILED DESCRIPTION:
Detailed Protocol

The following assessments will be undertaken by a consultant sports physician during the initial clinical examination:

* Hip joint range of motion (flexion, internal and external rotation)
* Flexion ADduction Internal Rotation (FADIR) and Flexion ABduction External Rotation (FABER) tests
* Squeeze tests (resisted adduction) at 90, 45 and 0 degrees were performed (SQ90°, SQ45° and SQ0° respectively)
* Resisted sit up
* Prone internal and external rotation
* Gaenslen's test
* Hip extension
* Femoral slump
* Thomas test
* Palpation of the adductor insertion to tubercle, pubic symphysis and superficial ring with resisted oblique sit up and deep ring scrotal invagination
* The crossover test Radiological examination will include magnetic resonance imaging of …..

Biomechanical testing involves the following progressive neuromuscular challenge tests which are undertaken after the clinical examination:

* Countermovement jump - Vertical jump as high as possible
* Single leg drop landing - Hop from a 30cm height onto one leg and hold the landing for 2sec
* Hurdle hop - Lateral hop over a 15cm hurdle followed by a hop back to the starting position and a hold for 2sec
* Change of direction cut - Sprint for 5 metres, make a 75 degree acute change of direction and sprint for a further five meters to the finish
* Indecision cut - Sprint for three meters then react to a light stimulus and make a 90 degree cut to the left or right for a further 1.5metres

Questionnaires

* Hip and groin outcome score (HAGOS)
* Marx activity rating scale

Physical therapy assessment:

* Single leg squat
* Straight leg raise
* Hip strength testing
* Hip range of motion
* Squeeze test
* Crossover test
* Linear running analysis

Rehabilitation Details

Movement Control Focusing on the deficits in large compound movement patterns evident during assessment as well as hip and trunk control deficits. High emphasis placed on the technical quality with which the sessions were carried out. Particular focus on pelvic control while improving sagittal and frontal plane hip and lumbopelvic control. Any symptoms during exercises indicates poor technique and the exercise will be reviewed and intensity reduced until appropriate technique achieved. The rep and set ranges reflected the emphasis on control while improving range at the thoracic spine, hip and ankle.

Strength-Power Double leg and single leg strength training carried out as necessary. Good form instructed throughout to ensure appropriate hip strategy especially under high load. Power work included single leg plyometric exercises to reduced ground contact and improve stiffness throughout the kinetic chain.

Linear Running Linear running drills focused on optimizing lumbo pelvic control in all three planes identified during assessment. Commence with wall drills and marching and skipping and progressing onto sled and harness drills which facilitate developing optimal posture with increased rate of force development and ground reaction forces to improve performance.

Multi Directional Multidirectional drills will be used to provide a neuromuscular challenge to the trunk on pelvis and hip control as well as optimizing foot position and the ability to control the centre of mass relative to the stance leg to reduce hip and pelvic overload and optimise cutting performance. Higher intensity cutting drills will be included as a progression once a painfree squeeze at 90 degrees has been achieved and symmetrical hip internal rotation bilaterally.

Conditioning With a view to ensuring all aspects of the athletes performance are addressed, conditioning will be carried out on a stationary bike to allow sufficient intensity without overloading the pubic/groin region. Sessions will be prescribed from Maximal Aerobic Power assessment on a wattbike and focused on alternate maximal and supramaximal sessions.

Hip and Groin Outcome Score (HAGOS) and MARX activity rating scale A HAGOS and MARX questionnaire will be completed by each groin patient on every visit -approximately every two weeks.

Patient Registry

Patient data will be inputted into iMedDoc medical data management software. Captured data will include:

Patient information - doubly de-identified patient code, electronic scan of consent form, anthropometric data, sport, playing position and playing level, time with pain, pain side or bilateral pain.

Sports medicine consultants findings - Diagnosis, magnetic resonance imaging findings, findings of clinical examination Physiotherapist's findings - clinical examination findings for initial test and post-rehabilitation HAGOS - hip and groin outcome score for initial test and throughout rehabilitation MARX activity rating scale - for initial test and throughout rehabilitation Magnetic resonance image files Quality assurance plan Weekly cross-checking will be undertaken by two members of staff to ensure data entered onto the registry is correct as per paper records and per acceptable ranges.

A six-monthly audit of the registry will be undertaken by external auditors (Dr Kieran Moran, Dublin City University and Dr Siobhan Strike, Roehampton University).

Registry standard operating procedures

Basic patient contact details are inputted by administration staff Patient consent form is uploaded to imeddoc software Doctors and physiotherapists input physical examination findings on imeddoc software HAGOS and Marx activity questionnaire are inputted by the patient using a tablet device. This data is uploaded to imeddoc automatically once questionnaire is completed.

Data is downloaded from imeddoc and placed into Microsoft excel. Patient name is de-identified.

Two researchers manage the registry updates and cross-check the data on a weekly basis. Where applicable paper records are checked to ensure the information submitted to the registry is complete and is within acceptable ranges.

A six-monthly audit of the registry will be undertaken by external auditors (Dr Kieran Moran, Dublin City University, Ireland and Dr Siobhan Strike, University of Roehampton, London).

Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect Suggested sample size = 600 Biomechanical clustering techniques (which will be used to describe the different biomechanical diagnoses that exist in AGP patients) require relatively large numbers of participants. Previous studies have utilised an n = 588 for this purpose (Sutherland and Davids), therefore it is hypothesised that 600 will be sufficient for such an analysis in the current study.

A sample size of n = 600 will allow a comprehensive examination of the clinical presentation of groin pain. Previous studies have only utilised up to 218 participants (Bradshaw et al 2008).

Finally, a sample size of 600 will be sufficient to account for drop out from the rehabilitation intervention. Drop out may be relatively high due to the regular physical therapy contact required (approximately every 2 weeks) despite the wide geographical spread of participants (throughout Ireland).

Registry Data Dictionary

Term Definition Rt Right Lt Left Dx Ant Plate Diagnosis of anterior plate pathology as a source of the groin pain Dx Hip Diagnosis of hip pathology as a source of the groin pain Dx Inguinal Diagnosis of inguinal ligament pathology as a source of the groin pain Dx Hip Flex Diagnosis of hip flexor pathology as a source of the groin pain Dx Labral Tear Diagnosis of hip labral tear pathology as a source of the groin pain Dx Apon Tear Diagnosis of pubic aponeurosis pathology as a source of the groin pain MRI BMO UNI Presence of bony oedema on magnetic resonance image - one side only MRI BMO BL Presence of bony oedema on magnetic resonance image - both sides MRI Rec Abd Ins Magnetic resonance image signal in the rectus abdominals insertion MRI Add Ins Magnetic resonance image signal in the adductor insertion MRI CAM Magnetic resonance image finding of a CAM hip impingement MRI FAI Magnetic resonance image finding of a femeroacetabular impingement MRI Apon Tear Magnetic resonance image finding of a aponeurosis tear Reduced Hip Flex Reduced hip flexion range of motion Reduced Hip IR Reduced hip internal range of motion Reduced Hip ER Reduced hip external range of motion FADIR Flexion, adduction and internal rotation symptomatic FABER Flexion, abduction and internal rotation symptomatic Squeeze 90 Squeeze test at 90 degrees is symptomatic Squeeze 45 Squeeze test at 45 degrees is symptomatic Squeeze 0 Straight leg squeeze test is symptomatic Thomas Thomas test symptomatic Mod Thom Modified Thomas test is symptomatic Res Leg Lift Resisted leg lift is symptomatic Adduct Tub Adductor tubercle is symptomatic on palpation Res Rot Resisted hip rotation is symptomatic Superf Inguin Ring Superficial inguinal ring symptomatic on palpation Rec Abd Insert Rectus abdominals insertion is symptomatic on palpation Deep Ring Deep inguinal ring is symptomatic on palpation Pubic Symp Pubic symphysis is symptomatic on palpation Slump Slump test positive SIJ Shear Sacro iliac joint shear is symptomatic Prone In/Et Rot Pronated internal/external hip rotation range of motion Femoral Slump Femoral slump test is positive Obs Lx Spine Observation of lumbar spine SL Squat Movement control in a single squat SL Bridge Lt Movement control in a single leg bridge Funct ASLR RT Functional active straight leg raise right Funct ASLR Lt Functional active straight leg raise right Res Hip Fle Resisted hip flexion strength test Hip Flex Hip flexion range of motion Hip IR Hip internal rotation range of motion Hip ER Hip external range of motion Prone IR Pronated hip internal rotation Short Hip FLex Short hip flexor range of motion Long Hip Flex Long hip flexor range of motion ASLR Active straight leg raise Crossover +ve Crossover test symptomatic Crossover -ve Crossover test non-symptomatic HAGOS Pain Pain score from the HAGOS questionnaire HAGOS Symptom Symptoms score from the HAGOS questionnaire HAGOS ADL Activities of daily living score from the HAGOS questionnaire HAGOS SportRec Sport and Recreation score from the HAGOS questionnaire HAGOS PA Physical activity score from the HAGOS questionnaire HAGOS QOL Quality of life score from the HAGOS questionnaire

Plan for missing data

Physical therapist completes a checklist once per week to flag missing data. This data is then completed from paper records.

Statistical analysis plan

Primary outcome measure (HAGOS) - Chi square test to examine changes in repeat HAGOS Secondary outcome measures (Kinetics and kinematics) - Repeated measures ANOVA to examine post-training changes in biomechanical variables Other outcome measures (Physical therapy measures) - Repeated measures ANOVA to examine post-training changes in physiotherapist measures

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of athletic groin pain
* Professional athlete in full time training with groin pain diagnosis

Exclusion Criteria:

* Post infective osteitis
* Bone tumour
* Acute injury

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 205 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Hip and groin outcome score (HAGOS) | Over the course of the rehabilitation time frame and one year and two years post initial consultation
  The HAGOS questionnaire is a validated tool (Thorborg et al. 2014; Thorborg et al. 2011) used to examine the impact of injury on physical function and to track symptoms at the time of diagnosis and as rehabilitation progresses.

SECONDARY OUTCOMES:
Kinetic and kinematic composite score | Following rehabilitation, an expected average of 10 weeks
  The post-training change in biomechanical measures following the intervention

OTHER OUTCOMES:
Hip range of movement | Following rehabilitation, an expected average of 10 weeks
  Post rehabilitation change in hip range as assessed by the physical therapist
Hip strength | Following rehabilitation, an expected average of 10 weeks
  Post rehabilitation change in hip strength as assessed by the physical therapist
Squeeze test | Following rehabilitation, an expected average of 10 weeks
  Using a pressure cuff, measure the pressure at which pain is felt
Cross-over test | Following rehabilitation, an expected average of 10 weeks
  Pain provocation test undertaken by physical therapist

CONTACTS AND LOCATIONS:
Overall Officials: Andy D Franklyn-Miller, MBBS, Study Director — Sports Surgery Clinic; Éanna C Falvey, MB, BCh, PhD, Study Director — Sports Surgery Clinic; Enda A King, BSc, MSc, Principal Investigator — Sports Surgery Clinic
Locations (1):
- Sports Surgery Clinic, Dublin, Leinster, Ireland

REFERENCES:
- [Background] Bradshaw CJ, Bundy M, Falvey E. The diagnosis of longstanding groin pain: a prospective clinical cohort study. Br J Sports Med. 2008 Oct;42(10):851-4. doi: 10.1136/bjsm.2007.039685. Epub 2008 Apr 1. PMID 18381826
- [Background] Holmich P, Thorborg K, Dehlendorff C, Krogsgaard K, Gluud C. Incidence and clinical presentation of groin injuries in sub-elite male soccer. Br J Sports Med. 2014 Aug;48(16):1245-50. doi: 10.1136/bjsports-2013-092627. Epub 2013 Aug 16. PMID 23956334
- [Background] Holmich P. Long-standing groin pain in sportspeople falls into three primary patterns, a "clinical entity" approach: a prospective study of 207 patients. Br J Sports Med. 2007 Apr;41(4):247-52; discussion 252. doi: 10.1136/bjsm.2006.033373. Epub 2007 Jan 29. PMID 17261557
- [Background] Holmich P, Uhrskou P, Ulnits L, Kanstrup IL, Nielsen MB, Bjerg AM, Krogsgaard K. Effectiveness of active physical training as treatment for long-standing adductor-related groin pain in athletes: randomised trial. Lancet. 1999 Feb 6;353(9151):439-43. doi: 10.1016/S0140-6736(98)03340-6. PMID 9989713
- [Background] Jardi J, Rodas G, Pedret C, Til L, Cusi M, Malliaropoulos N, Del Buono A, Maffulli N. Osteitis pubis: can early return to elite competition be contemplated? Transl Med UniSa. 2014 Apr 8;10:52-8. eCollection 2014 Sep. PMID 25147768
- [Background] Lovell G. The diagnosis of chronic groin pain in athletes: a review of 189 cases. Aust J Sci Med Sport. 1995 Sep;27(3):76-9. PMID 8599748
- [Background] Murphy JC, O'Malley E, Gissane C, Blake C. Incidence of injury in Gaelic football: a 4-year prospective study. Am J Sports Med. 2012 Sep;40(9):2113-20. doi: 10.1177/0363546512455315. Epub 2012 Aug 9. PMID 22879401
- [Background] Renstrom P, Peterson L. Groin injuries in athletes. Br J Sports Med. 1980 Mar;14(1):30-6. doi: 10.1136/bjsm.14.1.30. No abstract available. PMID 7378668
- [Background] Robinson P, Barron DA, Parsons W, Grainger AJ, Schilders EM, O'Connor PJ. Adductor-related groin pain in athletes: correlation of MR imaging with clinical findings. Skeletal Radiol. 2004 Aug;33(8):451-7. doi: 10.1007/s00256-004-0753-2. Epub 2004 Jun 29. PMID 15224172
- [Background] Serner A, van Eijck CH, Beumer BR, Holmich P, Weir A, de Vos RJ. Study quality on groin injury management remains low: a systematic review on treatment of groin pain in athletes. Br J Sports Med. 2015 Jun;49(12):813. doi: 10.1136/bjsports-2014-094256. Epub 2015 Jan 29. PMID 25633830
- [Background] Thorborg K, Branci S, Stensbirk F, Jensen J, Holmich P. Copenhagen hip and groin outcome score (HAGOS) in male soccer: reference values for hip and groin injury-free players. Br J Sports Med. 2014 Apr;48(7):557-9. doi: 10.1136/bjsports-2013-092607. Epub 2013 Jul 12. PMID 23850734
- [Background] Thorborg K, Bandholm T, Schick M, Jensen J, Holmich P. Hip strength assessment using handheld dynamometry is subject to intertester bias when testers are of different sex and strength. Scand J Med Sci Sports. 2013 Aug;23(4):487-93. doi: 10.1111/j.1600-0838.2011.01405.x. Epub 2011 Oct 28. PMID 22092308
- [Background] Walden M, Hagglund M, Ekstrand J. Football injuries during European Championships 2004-2005. Knee Surg Sports Traumatol Arthrosc. 2007 Sep;15(9):1155-62. doi: 10.1007/s00167-007-0290-3. Epub 2007 Mar 21. PMID 17375283
- [Derived] Franklyn-Miller A, Richter C, King E, Gore S, Moran K, Strike S, Falvey EC. Athletic groin pain (part 2): a prospective cohort study on the biomechanical evaluation of change of direction identifies three clusters of movement patterns. Br J Sports Med. 2017 Mar;51(5):460-468. doi: 10.1136/bjsports-2016-096050. Epub 2016 Oct 6. PMID 28209597
- [Derived] Falvey EC, King E, Kinsella S, Franklyn-Miller A. Athletic groin pain (part 1): a prospective anatomical diagnosis of 382 patients--clinical findings, MRI findings and patient-reported outcome measures at baseline. Br J Sports Med. 2016 Apr;50(7):423-30. doi: 10.1136/bjsports-2015-094912. Epub 2015 Nov 30. PMID 26626272